CLINICAL TRIAL: NCT06822335
Title: Evaluation of the Efficacy of Niacinamide a in the Management of Facial Post Inflammatory Hyperpigmentation (PIHP) Test Under Dermatological Control
Brief Title: Clinical Efficacy of the Product in the Management of Facial Post Inflammatory Hyperpigmentation (PIHP) Subjects
Status: Completed | Type: Observational
Sponsor: Cosmetique Active International (Industry)
Responsible Party: Sponsor
Other Study IDs: 2223CMCL076 _ LRP 22061
Record Dates: First submitted 2023-08-16; First posted 2025-02-12 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2023-08

CONDITIONS: Acne; Post-inflammatory Hyperpigmentation
MeSH Terms: conditions — Acne Vulgaris; Hyperpigmentation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Double-blind, randomized, clinical study is designed to evaluate the efficacy of Niacinamide A in the management of facial Post Inflammatory Hyper Pigmentation (PIHP) in healthy female and male subjects with moderate to severe PIHP due to acne, mild acne and (≤4) inflammatory lesions, its impact on skin lightening effect and lastly any associated benefits on skin quality.

DETAILED DESCRIPTION:
Primary objective To investigate the depigmenting effect of Niacinamide A in moderate to severe facial post inflammatory hyperpigmentation due to acne after a 12-week application period.

Secondary objectives

To evaluate any associated benefit of the product on skin condition and skin imperfection at different timepoints:

Product lightening efficacy using the Spectrocolorimeter. Evaluation of the global assessment evaluation for acne severity by the investigator using a 6 -point scale.

Counting of non-inflammatory and inflammatory lesions to access the change on the face.

Investigator scoring to assess the local intolerance (erythema, edema, dryness).

Subject scoring to assess the local intolerance(burning, stinging, itching and tingling sensations).

Subjective assessment of global tolerance of the product using a 4-point scale. Skin imaging analysis to assess the evaluation of the PIHP(darkness, size, number brown spots).

Evaluation of the mean darkness. Subjective evaluation of Global Assessment(SGA). Subject questionnaires to assess consumer perceived skin endpoints by filling in a cosmetic evaluation questionnaire and a stigmatization questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Female and male subjects aged between 18 - 50 years old.
* Subject of Fitzpatrick phototype III-VI.
* Subject must be willing and be able to comply with the study schedule, procedures, and restrictions.
* Subjects with moderate to severe scores (4-8) on mean darkness intensity.
* Subjects with moderate to severe PIHP due to acne (score PAPHI>10).
* Subjects with mild acne (GEA 2),
* Subjects having ≤ 4 inflammatory lesions total,
* Subjects showing understanding of the study procedures, restrictions, willingness to participate as evidenced by voluntary written informed consent.

Exclusion criteria

* Pregnant or intending to become pregnant during the study or breastfeeding or in menopause.
* Subjects under any hormonal therapy, such as contraceptive pills or androgen agonist/antagonist medications, within the last 3 months before Visit 1 or planning to start any therapy during the study.
* Subject with cutaneous pathology on the studied zone other than acne (eczema etc.).
* Use of topical or systemic treatment during the previous weeks liable to interfere with the assessment of the acceptability and efficacy of the studied products (according to the investigator's appreciation).
* Moderate to severe acne (GEA >2).
* Systemic treatment of retinoids during the six previous months of the study.
* Under retinoid treatment within the last 6 months, including Over. The Counter (OTC) and all derivates of retinoids (e.g., retinol, retinal, retinaldehyde, retinol esters, etc.).
* Under any acne medication (including oral medication/laser treatment) within the last 6 months.
* Subjects treated for PIHP within the past 3 months with either a cosmetic product or a drug.
* Subject with make-up products on the day of the visit at the center.
* Cosmetic product for non-comedogenicity within the last 2 weeks.
* History of skin cancer.
* History of abnormal response to sun.
* Presence of recent suntan (according to Investigator opinion) or photo-test marks.
* History of allergy, hypersensitivity, or any serious reaction to any cosmetic product.
* Any concomitant medical condition that may interfere with the study conduct in the opinion of the investigator.
* Having used within the month before inclusion any systemic medication for more than 5 consecutive days (e.g., steroidal, and non-steroidal anti-inflammatory drugs, corticoids, insulin, antihistamines, antihypertensive, antibiotics -e.g., quinolone, tetracycline, thiazides, fluoroquinolones-).
* Any subject who, in the judgment of the Investigator, should not participate in the study.
* Subject who cannot be contacted by telephone in case of emergency.
* Subject having participated within the 14 days before inclusion or currently participating in another clinical study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: female and male subjects with (Fitzpatrick phototype III-VI), aged between 18 and 50 years old, with moderate to severe PIHP due to acne (score PIHP > 10), with mild acne (GEA 2) and having inflammatory lesions (≤ 4 <10).
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2023-04-03 (Actual); Primary Completion 2023-08-07 (Actual); Study Completion 2023-08-08 (Actual)

PRIMARY OUTCOMES:
POST ACNE HYPERPIGMENTATION INDEX (PAHPI) | From baseline to Days 84
  The scoring will be performed by the Investigator with the PAHPI at etch visites. The score is composed by 3 parameters: Median Lesion size with 4 grades ( <3mm, 3-6mm, 7-10mm, >10 mm) , intensity with 3 grades ( slightly darker, Moderate darker, significant darker) and number of PIHP lesions with5 grades ( 01-15 lesions, 16-30 lesions, 31-45 lesions, 46-60 lésions, >60 lesions . The global score will be calculated (6 to 22).

SECONDARY OUTCOMES:
CLINICAL ASSESSMENT OF ACNE SEVERITY | From baseline to Days 84
  The dermatologist evaluates the acne severity according to the Global Acne Evaluation with the scale of 5 grades (0 Clear) to 5 ( Very severe)
Subject Global Assessment | From baseline to Days 84
  Global Evaluation with 6 grades ( -1, Worsered; 4 : Totally Cleared)

CONTACTS AND LOCATIONS:
Overall Officials: Gitanjali Gitanjali, MBBS, DDV, Principal Investigator — CIDP Ltée
Locations (1):
- CIDP Ltee, Port Louis, Mauritius

IPD SHARING:
Plan to Share IPD: No